CLINICAL TRIAL: NCT01331304
Title: Comparative Effectiveness of a Second Generation Antipsychotic Mood Stabilizer And a Classic Mood Stabilizer for Bipolar Disorder
Brief Title: Comparative Effectiveness Study for Bipolar Disorder
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Collaborators: Agency for Healthcare Research and Quality (AHRQ) (U.S. Federal Agency)
Responsible Party: Principal Investigator, Andrew A. Nierenberg, MD, Director of Research, Bipolar Clinic and Research Program, Massachusetts General Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2010P001442; R01HS019371-01 (AHRQ)
Record Dates: First submitted 2011-04-06; First posted 2011-04-08 (Estimated); Results first posted 2014-06-04 (Estimated); Last update posted 2018-04-26 (Actual); Status verified 2018-03

CONDITIONS: Bipolar Disorder
Keywords: Bipolar disorder; Comparative effectiveness trial; Lithium; Quetiapine
MeSH Terms: conditions — Bipolar Disorder | interventions — Lithium; Lithium Carbonate; Quetiapine Fumarate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Li + APT (Other): Study participants will take lithium in addition to any other medications recommended by the study physician.
  Interventions: Drug: Lithium
- QTP + APT (Other): Study participants will take quetiapine in addition to any other medications recommended by the study physician.
  Interventions: Drug: Quetiapine

INTERVENTIONS:
Drug: Lithium — 600-900mg per day over 6 months
  Other Names: Lithoboid, Eskalith
  Arms: Li + APT
Drug: Quetiapine — 100-800mg a day over 6 months
  Other Names: Seroquel
  Arms: QTP + APT

SUMMARY:
The purpose of this study is to compare the effectiveness of lithium and quetiapine for the treatment of individuals with bipolar disorder.

DETAILED DESCRIPTION:
Mood stabilizers, medications that prevent future mood episodes, are the foundation for treatment of bipolar disorder. While all published bipolar disorder treatment guidelines recommend that pharmacotherapy should include mood stabilizers for long-term maintenance treatment, no randomized comparative effectiveness studies have examined the real-world advantages and disadvantages of the newer second generation antipsychotic (SGA) mood stabilizers compared to the classic mood stabilizers, such as lithium (Li). No studies have looked at the effectiveness of SGAs compared to mood stabilizers when used in the context of other medications required to manage bipolar patients, since bipolar disorder patients take a median of 3 medications for optimal outcomes. Quetiapine (QTP) is the most extensively studied, broadly efficacious and the most widely prescribed SGA for bipolar disorder. The classic mood stabilizer Li has the largest evidence base for treating bipolar disorder, but has been largely supplanted by the SGAs.

Thus, this study compares symptomatic benefits and adverse effect burden between a QTP foundation with adjunctive personalized treatments (QTP+APT) and a mood stabilizer foundation consisting of Li with APT (Li+APT). APT will include any other medication needed with the following exceptions: the QTP+APT cannot receive Li and the Li+APT group cannot receive an antipsychotic. If, however, participants clinically require a switch to, or the addition of any other SGA or mood stabilizer, then those medications can be added as a rescue strategy that will be carefully recorded. Consistent with an effectiveness trial, participants will be able to continue in the study if they require a rescue treatment. The specific plan is a randomized, open, two arm, comparative effectiveness study of QTP+APT vs. Li+APT treatment for 6 months across 10 sites.

In summary, this comparative effectiveness study compares fundamentally different acute and continuation treatments for bipolar disorder. The investigators address the key question of whether to use a prototypical mood stabilizing SGA (i.e., QTP) or the classical mood stabilizer Li as the foundational treatment in the context of other necessary adjunctive personalized treatments (APT).

ELIGIBILITY:
Inclusion Criteria:

1. Meets DSM-IV criteria for BD I or II, which is the primary focus of treatment
2. Able to give written informed consent
3. Age > to 18 years and < 68 years
4. Women of child bearing potential must agree to use adequate contraception (e.g. oral contraceptives, intrauterine device, barrier methods, or total abstinence from intercourse; Depo Provera is acceptable if it is started 3 months prior to enrollment), inform their doctor at the earliest possible time of their plans to conceive, and to understand the risks of lithium and other study treatments to the fetus and infant
5. Currently symptomatic, as defined as a Clinical Global Impression - Bipolar Disorder Overall Severity (CGI-BP-S) score of at least 3 (mild)
6. If currently taking an SGA, participants would be required to be willing to either discontinue or switch to QTP
7. Willing to be randomized to either QTP+APT or Li+APT.

Exclusion Criteria:

1. Unwilling or unable to comply with study requirements
2. If maintained on thyroid medication must be euthyroid for at least 1 month before Visit 1
3. Patients who have had intolerable side effects with QTP or Li
4. Patients whose clinical status requires inpatient care
5. Drug/alcohol dependence within the past 30 days
6. Pregnancy as determined by urine pregnancy test or breastfeeding
7. History of nonresponse to Li at a serum level of ≥ 1.0 mEq/L ≥ 8 weeks
8. History of nonresponse to QTP at doses of at least 600 mg ≥ 8 weeks.

Ages: 18 Years to 68 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 482 (Actual)
Dates: Start 2010-09; Primary Completion 2013-04 (Actual); Study Completion 2013-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Andrew A Nierenberg, MD, Principal Investigator — Massachusetts General Hospital
Locations (11):
- United States (11):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - Stanford University School of Medicine, Stanford, California
  - Massachusetts General Hospital, Boston, Massachusetts
  - University of Michigan, Ann Arbor, Michigan
  - Weill Cornell Medical College, New York, New York
  - Case Western Reserve University School of Medicine, Cleveland, Ohio
  - The Lindner Center of HOPE, Mason, Ohio
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania
  - Vanderbilt University, Nashville, Tennessee
  - The University of Texas Health Science Center, San Antonio, Texas

REFERENCES:
- [Derived] Sylvia LG, Montana RE, Deckersbach T, Thase ME, Tohen M, Reilly-Harrington N, McInnis MG, Kocsis JH, Bowden C, Calabrese J, Gao K, Ketter T, Shelton RC, McElroy SL, Friedman ES, Rabideau DJ, Nierenberg AA. Poor quality of life and functioning in bipolar disorder. Int J Bipolar Disord. 2017 Dec;5(1):10. doi: 10.1186/s40345-017-0078-4. Epub 2017 Mar 27. PMID 28188565
- [Derived] Deckersbach T, Nierenberg AA, McInnis MG, Salcedo S, Bernstein EE, Kemp DE, Shelton RC, McElroy SL, Sylvia LG, Kocsis JH, Bobo WV, Friedman ES, Singh V, Tohen M, Bowden CL, Ketter TA, Calabrese JR, Thase ME, Reilly-Harrington NA, Rabideau DJ, Kinrys G, Kamali M. Baseline disability and poor functioning in bipolar disorder predict worse outcomes: results from the Bipolar CHOICE study. J Clin Psychiatry. 2016 Jan;77(1):100-8. doi: 10.4088/JCP.14m09210. PMID 26845265
- [Derived] Nierenberg AA, McElroy SL, Friedman ES, Ketter TA, Shelton RC, Deckersbach T, McInnis MG, Bowden CL, Tohen M, Kocsis JH, Calabrese JR, Kinrys G, Bobo WV, Singh V, Kamali M, Kemp D, Brody B, Reilly-Harrington NA, Sylvia LG, Shesler LW, Bernstein EE, Schoenfeld D, Rabideau DJ, Leon AC, Faraone S, Thase ME. Bipolar CHOICE (Clinical Health Outcomes Initiative in Comparative Effectiveness): a pragmatic 6-month trial of lithium versus quetiapine for bipolar disorder. J Clin Psychiatry. 2016 Jan;77(1):90-9. doi: 10.4088/JCP.14m09349. PMID 26845264
- [Derived] Bobo WV, Reilly-Harrington NA, Ketter TA, Brody BD, Kinrys G, Kemp DE, Shelton RC, McElroy SL, Sylvia LG, Kocsis JH, McInnis MG, Friedman ES, Singh V, Tohen M, Bowden CL, Deckersbach T, Calabrese JR, Thase ME, Nierenberg AA, Rabideau DJ, Schoenfeld DA, Faraone SV, Kamali M. Complexity of illness and adjunctive benzodiazepine use in outpatients with bipolar I or II disorder: results from the Bipolar CHOICE study. J Clin Psychopharmacol. 2015 Feb;35(1):68-74. doi: 10.1097/JCP.0000000000000257. PMID 25514063

RESULTS

PARTICIPANT FLOW:
Groups:
- Li + APT: Study participants will take lithium in addition to any other medications recommended by the study physician.
  Lithium: 600-1200mg per day over 6 months
Period: Overall Study
Arm/Group | Li + APT | QTP + APT
Started | 240 | 242
Completed | 182 | 182
Not Completed | 58 | 60

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Li + APT | QTP + APT | Total
Number analyzed (Participants) | 240 | 242 | 482
Age, Continuous [Mean (Standard Deviation); unit: Years] | 38.6 (12.1) | 39.1 (12.2) | 38.9 (12.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 140 | 143 | 283
  Male | 100 | 99 | 199
Region of Enrollment [Number; unit: participants]
  United States | 240 | 242 | 482

OUTCOME MEASURES:

1. Primary Outcome: Clinical Global Impression-Efficacy Index (CGI-EI)
Description: The CGI-EI integrates benefits and harms and yields a score that can be compared across interventions. It is made up of 2 subscales: therapeutic effects and side effects. Each rating is on a scale from 1 to 4. To combine these two subscales into the CGI-EI we report as our primary outcome, we subtracted the side effects subscale from the therapeutic effects subscale. Thus, the CGI-EI we report ranges the integers from -3 to +3 (i.e. possible scores are -3,-2,-1,0,1,2,3). A score of -3 is the most burdensome side effect score (4) and the least therapeutic effect score (1) and a score of +3 is the least burdensome side effect score (1) and the highest therapeutic effect score (4). Higher CGI-EI signifies better outcome (minimal side effects, maximal therapeutic effect). Lower CGI-EI signifies worse outcome (maximal side effects, minimal therapeutic effect).To compute CGI-EI score, we subtract the side effect score from the therapeutic effect score.
Time Frame: Average 6 month score minus Average baseline score
Measure: Mean (95% Confidence Interval); unit: Units on the scale
Arm/Group | Li + APT | QTP + APT
Number analyzed (Participants) | 240 | 242
Units on the scale | 1.58 [1.32 to 1.84] | 1.52 [1.26 to 1.78]
Statistical Analysis 1: Comparison: Li + APT vs QTP + APT; For the first co-primary aim, mixed-effects linear regression analyses compared the two intervention groups on the repeated assessments of the CGI-EI over 6 months; Test type: Superiority or Other; p = 0.59, Mixed Models Analysis — Because this study has co-primary outcomes (CGI-EI and NCAs), the analyses of the treatment effect in the two primary hypotheses each involved a two-tailed alpha-level of 0.025

2. Primary Outcome: Necessary Clinical Adjustments
Description: Necessary Clinical Adjustment (NCA): The Medication Recommendation Tracking Form was developed and successfully implemented in a previous study to capture recommended medication changes at each study visit 17. Clinicians record dosage changes, missed doses, new medications added or discontinued, and specify the reason for each change. Any change in psychotropic medications, or medications used to treat side effects, is coded along with the reason for the change. NCAs include those changes made for lack of effectiveness or intolerance, but not changes for planned dose titrations.
Time Frame: 6 Months
Measure: Mean (Standard Deviation); unit: Mean NCAs per month
Arm/Group | Li + APT | QTP + APT
Number analyzed (Participants) | 240 | 242
Mean NCAs per month | .8 (.8) | .9 (1.0)
Statistical Analysis 1: Comparison: Li + APT vs QTP + APT; For the second co-primary, patient monthly rates of NCAs (determined by dividing total number of NCAs during follow-up by the length of follow-up - to account for attrition and resulting differential exposure time) for treatment groups were compared using a Wilcoxon rank-sum test; Test type: Superiority or Other; p = 0.118, Wilcoxon (Mann-Whitney)

3. Secondary Outcome: Risk of Cardiovascular Disease - Framingham Risk Score
Description: The Framingham risk score captures the classic risk factors for cardiovascular disease, including age, sex, systolic blood pressure, total and high density lipoprotein cholesterol, diabetes mellitus, and smoking. The Framingham risk score is used as a simple predictive tool to determine 10-year (short term) risk for developing cardiovascular disease (CHD), with higher scores indicating higher risk. Established benchmarks exist for scores from 0 to 25--though it can exceed this value--that are meant to translate to the probability of developing heart disease.
Time Frame: Average baseline score minus Average 6 month score
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Li + APT | QTP + APT
Number analyzed (Participants) | 240 | 242
units on a scale | -0.26 [-0.66 to 0.14] | 0.17 [-0.21 to 0.54]
Statistical Analysis 1: Comparison: Li + APT vs QTP + APT; Mixed-effects linear regression analyses compared the two intervention groups on the repeated collection of measures relevant to calculation of the Framingham Risk Score over 6 months; Test type: Superiority; p = 0.11, Mixed Models Analysis — Analysis of this secondary outcome was not corrected for multiple comparisons. Therefore, the a priori threshold for statistical significance was set at 0.05

4. Secondary Outcome: Longitudinal Interval Follow up Evaluation Range of Impaired Functioning Tool (LIFE-RIFT)
Description: The LIFE-RIFT asses the extent to which psychopathology has impacted current functioning in work, household chores, interpersonal relationships with partner, family, and friends, recreational activities, and life, satisfaction, leisure activities and social relationships. Summary scores can range from 4 to 20, with higher scores indicating greater functional impairment.
Time Frame: Average baseline score minus Average 6-month score
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Li + APT | QTP + APT
Number analyzed (Participants) | 240 | 242
units on a scale | -3.74 [-4.29 to -3.19] | -3.61 [-4.15 to -3.07]
Statistical Analysis 1: Comparison: Li + APT vs QTP + APT; Mixed-effects linear regression analyses compared the two intervention groups on the repeated assessment of the LIFE-RIFT over 6 months; Test type: Superiority; p = 0.70, Mixed Models Analysis — [p-value comment as in outcome 3, analysis 1]

ADVERSE EVENTS:
Time Frame: Six months
Arm/Group | Li + APT | QTP + APT
Serious Adverse Events (participants affected / at risk) | 36/240 | 27/242
Other Adverse Events (participants affected / at risk) | 210/240 | 221/242
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Li + APT (N=240) | QTP + APT (N=242)
Pregnancy (Pregnancy, puerperium and perinatal conditions) | 3 (3) | 1 (1)
Psychiatric Hospitalization (Psychiatric disorders) | 18 (23) | 14 (19)
Car/Bike Accident (Injury, poisoning and procedural complications) | 2 (2) | 1 (1)
Suicide (Psychiatric disorders) | 1 (1) | 0 (0)
Death (Cardiac disorders) | 1 (1) | 0 (0)
Laparoscopic Cholecystectomy (Surgical and medical procedures) | 1 (1) | 0 (0)
Alcoholism Treatment (General disorders) | 1 (1) | 0 (0)
Gastrointestinal Issues (Gastrointestinal disorders) | 2 (2) | 0 (0)
Kidney Infection (Renal and urinary disorders) | 1 (1) | 0 (0)
Heroin Overdose (General disorders) | 1 (1) | 0 (0)
Eczema Outbreak (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Hospitalization reason unknown (General disorders) | 0 (0) | 1 (1) — Hospitalization reason unknown; unable to re-contact study participant
Broken Bones (Injury, poisoning and procedural complications) | 0 (0) | 2 (2)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 2 (2)
Flu Hospitalization (Infections and infestations) | 0 (0) | 1 (1)
Extreme Sedation Hospitalization (General disorders) | 0 (0) | 1 (1)
Muscle Spasms Hospitalization (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Biliary Cirrhosis (Hepatobiliary disorders) | 1 (1) | 0 (0)
Study Medication Overdose (General disorders) | 1 (1) | 2 (2)
Pseudoseizure (Nervous system disorders) | 1 (1) | 0 (0)
Cyst (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Staph Infection (Infections and infestations) | 0 (0) | 1 (1)
Dizziness (General disorders) | 1 (1) | 0 (0) — Adverse reaction to study medication: dizziness, disturbance in gait
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Li + APT (N=240) | QTP + APT (N=242)
Excessive sleepiness/daytime somnolence (General disorders) | 68 (96) | 186 (249)
Headache (Nervous system disorders) | 48 (61) | 33 (43)
Dry Mouth (General disorders) | 29 (32) | 51 (58)
Nausea (Gastrointestinal disorders) | 58 (70) | 15 (17)
Increased Weight (General disorders) | 25 (31) | 45 (55)
Tremor (Musculoskeletal and connective tissue disorders) | 63 (69) | 13 (13)
Increased Appetite (General disorders) | 20 (22) | 55 (56)
Memory/concentration problems (Nervous system disorders) | 27 (32) | 21 (25)
Dizziness/Lightheaded (Nervous system disorders) | 21 (24) | 23 (30)
Upset stomach/stomach pain/bloating (Gastrointestinal disorders) | 31 (36) | 12 (13)
Diarrhea (Gastrointestinal disorders) | 32 (38) | 7 (10)
Constipation (Gastrointestinal disorders) | 19 (23) | 22 (23)
Increased Thirst (General disorders) | 29 (32) | 4 (4)
Increased Urinary Frequency (Renal and urinary disorders) | 32 (33) | 2 (3)
Stiffness/muscle aches (Musculoskeletal and connective tissue disorders) | 13 (14) | 14 (14)
Weakness/muscle fatigue (Musculoskeletal and connective tissue disorders) | 11 (12) | 14 (15)
Restless/fidgety (akathisia) (General disorders) | 7 (7) | 15 (17)
Respiratory infection or other cold-like symptoms (Respiratory, thoracic and mediastinal disorders) | 12 (12) | 12 (12)
Muscle twitching (myoclonus) (Musculoskeletal and connective tissue disorders) | 6 (6) | 14 (14)
Hair Loss (Skin and subcutaneous tissue disorders) | 16 (16) | 4 (4)
Blurred Vision (Eye disorders) | 12 (15) | 6 (7)
Insomnia (General disorders) | 12 (12) | 5 (7)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No